CLINICAL TRIAL: NCT00575432
Title: Evaluation of Kidney Function by Multi-modal Magnetic Resonance Imaging and Spectroscopy in Renal Transplantation and Kidney Disease
Brief Title: Evaluation of Kidney Function by Multi-modal Magnetic Resonance Imaging and Spectroscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: KEK 213/04; 1066
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Kidney Transplantation; Urinary Calculi
Keywords: magnetic resonance imaging; renal function; renal transplant; urinary calculi; healthy controls; kidney
MeSH Terms: conditions — Urinary Calculi | interventions — Diffusion Tensor Imaging; Treatment Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Radiation: diffusion MRI; Radiation: BOLD MRI; Other: Clinical Outcome

INTERVENTIONS:
Radiation: diffusion MRI — diffusion MRI
Radiation: BOLD MRI — BOLD MRI
Other: Clinical Outcome — Clinical outcome

SUMMARY:
Multimodal functional magnetic resonance (MR) methods, including MR diffusion, Blood-Oxygenation Level Dependent (BOLD) imaging and MR spectroscopy may provide complementary information about the functional status of a kidney. The researchers hypothesize that these non-invasive methods correlate with histology as "gold standard" and compete favorably with conventional in part invasive evaluation methods, and thus provide specific and early detection of kidney diseases of various etiologies, drug toxicity, or renal allograft dysfunction.

DETAILED DESCRIPTION:
Early and specific detection of dysfunction in kidney diseases and differential diagnosis of potential complications in the renal allograft are fundamental to initiate appropriate treatment. In addition, determination of renal function may reveal physiological mechanisms that may prove useful for future therapeutic procedures. Currently, used methods to access renal function like ultrasound, radionuclide imaging, and laboratory methods have several disadvantages, as they are nonspecific, require radioactive contrast agents or are limited in spatial information. Therefore, alternative non-invasive methods to detect early morphological and functional changes are required. Recently, a variety of very promising advanced magnetic resonance imaging (MRI) methods have evolved to obtain functional information of different organs. These methods include MR angiography, diffusion, perfusion and Blood-Oxygenation Level Dependent (BOLD) imaging. In addition to MRI, MR spectroscopy (MRS) provides renal functional information. In abdominal organs like the kidney, respiratory, and cardiac motion and susceptibility artifacts have limited the use of these functional MR methods for clinical applications. However, this may be overcome with the advent of greatly enhanced hardware, allowing very fast imaging times. Besides these in vivo techniques, novel processing algorithms for complex ex vivo MR spectra of body fluids have emerged recently. These methods, labeled "Metabonomics", access renal function by obtaining metabolic profiles that are indicative for renal dysfunction.

The researchers hypothesize that these non-invasive methods correlate with histology as "gold standard" and compete favorably with conventional in part invasive evaluation methods, and thus provide specific and early detection of kidney diseases of various etiologies, drug toxicity or renal allograft dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 16 years
* Male or female
* Signed consensus report to the study

Exclusion Criteria:

* History of allergy to contrast media
* Pregnancy
* Contraindication for MR examination: Content of electronic devices in the body of the subject (i.e. pacemaker of heart, implanted insulin pump, nerve stimulator, or similar medical devices), content of metallic foreign bodies or metal-pieces (without amalgam filling), claustrophobia
* Back or other problems that don't allow motionless lying for 75 minutes
* Missing signed consensus report to the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Kidney diseases and Renal Allografts
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2004-11; Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of functional MR parameters with histology results as "gold standard" or with final clinical outcome | 6 months

SECONDARY OUTCOMES:
Correlation with clinical results, laboratory results (e.g. GFR, serum-creatinine levels), results from other imaging procedures, correlation within MR parameters (e.g. in vivo metabolites vs. in vitro (from urine) metabolites, oxygenation vs. diffusion) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Harriet C Thoeny, MD, Principal Investigator — Institute of Radiology, University of Bern; Peter Vermathen, PhD, Principal Investigator — University Bern, Dept.Clinical Research
Locations (1):
- Department of Diagnostic and Interventional Neuroradiology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mani LY, Seif M, Nikles F, Tshering Vogel DW, Diserens G, Martirosian P, Burnier M, Vogt B, Vermathen P. Hip Position Acutely Affects Oxygenation and Perfusion of Kidney Grafts as Measured by Functional Magnetic Resonance Imaging Methods-The Bent Knee Study. Front Med (Lausanne). 2021 Aug 10;8:697055. doi: 10.3389/fmed.2021.697055. eCollection 2021. PMID 34447762
- [Background] Mani LY, Cotting J, Vogt B, Eisenberger U, Vermathen P. Influence of Immunosuppressive Regimen on Diffusivity and Oxygenation of Kidney Transplants-Analysis of Functional MRI Data from the Randomized ZEUS Trial. J Clin Med. 2022 Jun 8;11(12):3284. doi: 10.3390/jcm11123284. PMID 35743353
- [Result] Giannarini G, Kessler TM, Roth B, Vermathen P, Thoeny HC. Functional multiparametric magnetic resonance imaging of the kidneys using blood oxygen level dependent and diffusion-weighted sequences. J Urol. 2014 Aug;192(2):434-9. doi: 10.1016/j.juro.2014.02.048. Epub 2014 Feb 25. PMID 24582541
- [Result] Eisenberger U, Binser T, Thoeny HC, Boesch C, Frey FJ, Vermathen P. Living renal allograft transplantation: diffusion-weighted MR imaging in longitudinal follow-up of the donated and the remaining kidney. Radiology. 2014 Mar;270(3):800-8. doi: 10.1148/radiol.13122588. Epub 2013 Nov 13. PMID 24475796
- [Result] Binser T, Thoeny HC, Eisenberger U, Stemmer A, Boesch C, Vermathen P. Comparison of physiological triggering schemes for diffusion-weighted magnetic resonance imaging in kidneys. J Magn Reson Imaging. 2010 May;31(5):1144-50. doi: 10.1002/jmri.22156. PMID 20432350
- [Result] Eisenberger U, Thoeny HC, Binser T, Gugger M, Frey FJ, Boesch C, Vermathen P. Evaluation of renal allograft function early after transplantation with diffusion-weighted MR imaging. Eur Radiol. 2010 Jun;20(6):1374-83. doi: 10.1007/s00330-009-1679-9. Epub 2009 Dec 16. PMID 20013274
- [Result] Thoeny HC, Kessler TM, Simon-Zoula S, De Keyzer F, Mohaupt M, Studer UE, Vermathen P. Renal oxygenation changes during acute unilateral ureteral obstruction: assessment with blood oxygen level-dependent mr imaging--initial experience. Radiology. 2008 Jun;247(3):754-61. doi: 10.1148/radiol.2473070877. Epub 2008 Apr 10. PMID 18403623
- [Result] Thoeny HC, Zumstein D, Simon-Zoula S, Eisenberger U, De Keyzer F, Hofmann L, Vock P, Boesch C, Frey FJ, Vermathen P. Functional evaluation of transplanted kidneys with diffusion-weighted and BOLD MR imaging: initial experience. Radiology. 2006 Dec;241(3):812-21. doi: 10.1148/radiol.2413060103. PMID 17114628
- [Result] Thoeny HC, Binser T, Roth B, Kessler TM, Vermathen P. Noninvasive assessment of acute ureteral obstruction with diffusion-weighted MR imaging: a prospective study. Radiology. 2009 Sep;252(3):721-8. doi: 10.1148/radiol.2523082090. PMID 19567650
- [Result] Seif M, Lu H, Boesch C, Reyes M, Vermathen P. Image registration for triggered and non-triggered DTI of the human kidney: reduced variability of diffusion parameter estimation. J Magn Reson Imaging. 2015 May;41(5):1228-35. doi: 10.1002/jmri.24671. Epub 2014 Jun 25. PMID 24962556
- [Result] Seif M, Eisenberger U, Binser T, Thoeny HC, Krauer F, Rusch A, Boesch C, Vogt B, Vermathen P. Renal Blood Oxygenation Level-dependent Imaging in Longitudinal Follow-up of Donated and Remaining Kidneys. Radiology. 2016 Jun;279(3):795-804. doi: 10.1148/radiol.2015150370. Epub 2016 Jan 8. PMID 26744926
- [Result] Seif M, Mani LY, Lu H, Boesch C, Reyes M, Vogt B, Vermathen P. Diffusion tensor imaging of the human kidney: Does image registration permit scanning without respiratory triggering? J Magn Reson Imaging. 2016 Aug;44(2):327-34. doi: 10.1002/jmri.25176. Epub 2016 Feb 12. PMID 26871263